CLINICAL TRIAL: NCT01495676
Title: A Randomized Phase II Trial Evaluating an Organ-conserving Strategy With Radiotherapy + CDDP + Gemcitabine vs Radiotherapy + CDDP in Muscle-infiltrative Bladder Cancer
Brief Title: A Phase II Trial Evaluating an Organ-conserving Strategy by Radiochemotherapy for Muscle-infiltrative Bladder Cancer
Acronym: GETUGV04
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETUG V04; 2011-000408-17 (EudraCT Number)
Record Dates: First submitted 2011-12-14; First posted 2011-12-20 (Estimated); Results first posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-07

CONDITIONS: Infiltrating Bladder Urothelial Carcinoma
Keywords: Bladder cancer; Organ-conserving strategy; Radiochemotherapy; non metastatic
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Radiation; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiotherapy + cisplatin (Active Comparator)
  Interventions: Other: Radiation + cisplatin
- Radiotherapy + cisplatin + gemcitabine (Experimental)
  Interventions: Other: Radiation + cisplatin + gemcitabine

INTERVENTIONS:
Other: Radiation + cisplatin — RT will encompass bilateral internal and external iliac lymph nodes at a dose of 45 Gy and the bladder up to 63 Gy. Fractionation will be 1.8 Gy per fraction.
  Cisplatin: 20 mg/m2/day through continuous iv perfusion for 4 consecutive days, from D2 to D5 and from D23 to D26 for the first part of the treatment, then from D2 to D5 if an additional treatment is decided.
  A cystoscopy with a transurethral resection will be performed 3 weeks after the last day of the first part of radio-chemotherapy.
  * In the absence of tumor cells, the 2nd part will start on the 4th week or at latest on the 5th week after the last day of the 1st part of radio-chemotherapy.
  * In case of a microscopic tumor residue or of a local tumor progression, operability will be re-evaluated in view of a radical cystectomy and the patient will exit the study.
  Arms: Radiotherapy + cisplatin
Other: Radiation + cisplatin + gemcitabine — Radiotherapy will encompass bilateral internal and external iliac lymph nodes at a dose of 45 Gy and the bladder up to 63 Gy. Fractionation will be 1.8 Gy per fraction.
  Cisplatin: 20 mg/m2/day through continuous iv perfusion for 4 consecutive days, from D2 to D5 and from D23 to D26 for the first part of the treatment, then from D2 to D5 for the second part of the treatment if an additional treatment is decided.
  Gemcitabine: iv injection for 30 minutes, twice a week at a dose of 25 mg/m2 on days 2, 5, 9, 12, 16, 19, 23, 26, 30, and 33 for the 1st part of treatment, then on days 2, 5, 9, and 12 for the 2nd part of treatment if an additional treatment is decided (cystoscopy with a transurethral resection). RT will be delivered between 2 and 6 hours after completion of the gemcitabine injection.
  Arms: Radiotherapy + cisplatin + gemcitabine

SUMMARY:
If radical cystectomy remains the standard of care for muscle invasive bladder cancer, consequences of this surgical procedure are often harsh. Over the past years, concurrent chemo-radiotherapy has imposed itself as an alternative treatment. Published data on concomitant radiochemotherapy (radiotherapy/cisplatin or radiotherapy/cisplatin/5-fluorouracil combinations) showed local control rates with bladder preservation at 5 years ranging from 40% to 65% according to the disease stage, and overall survival probabilities ranging from 40% to 50% at 5 years. In order to improve local and systemic prognosis, evaluation of other chemotherapy agents with higher radiosensitizing effect, such as gemcitabine, is justified. Gemcitabine possesses its own anti-cancer activities on urothelial diseases and has a synergetic activity with cisplatin. The investigators completed a monocenter phase I study combining radiotherapy, cisplatin, and twice-weekly gemcitabine, and determined a recommended dose of gemcitabine 25 mg/m². The objective of the present study is to evaluate the combination of radiotherapy + cisplatin + gemcitabine in terms of disease-free survival in non metastatic muscle invasive urothelial cancer patients.

DETAILED DESCRIPTION:
The objective of the present study is to evaluate the combination of radiotherapy + cisplatin + gemcitabine in terms of disease-free survival in non metastatic muscle invasive urothelial cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Muscle invasive urothelial cancer (front line or following the progression of a superficial tumor), pT2-pT3 stage without lymphatic impairment (N0) and without detectable metastases (M0). An optimal macroscopic resection (TURB) have to be performed
* The proof of invasive tumor to the muscle should be brought by a transurethral resection under anaesthesia less than 8 weeks before or, in the absence, by superficial biopsies and formal imaging. Multiples biopsies in the bladder must also be performed.
* Age ≥ 18 years
* Life expectancy ≥ 6 months
* Kanorfsky index ≥ 70 % (WHO 0, 1, 2)
* Biological criteria: neutrophils ≥ 1500/mm3, Platelets ≥ 100 000/mm3, haemoglobin ≥ 10 g/dl, creatinine clearance > 60 ml/mn
* No distant metastases (Thorax, abdomen, and pelvic CT-scan, bone scan)
* Efficient contraception for premenopausal women, maintained during the whole treatment and up to two months after the completion of radiotherapy.
* No radiotherapy or chemotherapy history except for in situ bladder lesions.
* No carcinological history except for non melanoma skin tumours, in situ uterine cervix cancer
* No contraindication to gemcitabine or cisplatin.
* No contraindication to radiotherapy
* Information letter and informed consent signed
* Patient covered by social security

Exclusion Criteria:

* Bladder tumors without any muscle infiltration
* Epidermoid carcinoma or adenocarcinoma
* Distance metastases or extrapelvic node positivity
* Severe digestive history (ulcerative colitis, complicated diverticulitis)
* Pregnancy and breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-07-06 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2024-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Azria David, MD, Study Chair — ICM Val d'Aurelle
Locations (12):
- France (12):
  - Institut Bergonié, Bordeaux
  - Centre Francois Baclesse, Caen
  - Hopital Henri Mondor, Créteil
  - CRLC GF Leclerc, Dijon
  - CRLC Val d'Aurelle-Paul Lamarque, Montpellier
  - Centre azuréen de Cancérologie, Mougins
  - Centre Antoine Lacassagne, Nice
  - Hopital saint Louis, Paris
  - HEGP, Paris
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Clinique Patseur, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No
Individual data are listed in the form of datalistings (lists by chapter) and "patient profile" (summary of main data per patient). The database is frozen for validated data. This basic freezing is done by the dated copy of the database and then by a selection of observations meeting the criteria. This process is repeated until the complete recovery of the validated data.

REFERENCES:
- [Background] Azria D, Jacot W, Prost P, Culine S, Ychou M, Lemanski C, Dubois JB. [Gemcitabine and ionizing radiations: radiosensitization or radio-chemotherapy combination]. Bull Cancer. 2002 Apr;89(4):369-79. French. PMID 12016038
- [Background] Caffo O, Fellin G, Graffer U, Valduga F, Bolner A, Luciani L, Tomio L, Galligioni E. Phase I study of gemcitabine and radiotherapy plus cisplatin after transurethral resection as conservative treatment for infiltrating bladder cancer. Int J Radiat Oncol Biol Phys. 2003 Dec 1;57(5):1310-6. doi: 10.1016/s0360-3016(03)00763-6. PMID 14630267
- [Background] Chauvet B, Brewer Y, Felix-Faure C, Davin JL, Choquenet C, Reboul F. Concurrent cisplatin and radiotherapy for patients with muscle invasive bladder cancer who are not candidates for radical cystectomy. J Urol. 1996 Oct;156(4):1258-62. PMID 8808849
- [Background] Chauvet B, Davin JL, Alfonsi M, Berger C, Vincent P, Reboul F. [Conservative treatment of bladder cancers with radiotherapy and concurrent chemotherapy: results and perspectives]. Cancer Radiother. 1998 Sep-Oct;2(5):499-504. doi: 10.1016/s1278-3218(98)80058-9. French. PMID 9868392
- [Background] Choudhury A, Swindell R, Logue JP, Elliott PA, Livsey JE, Wise M, Symonds P, Wylie JP, Ramani V, Sangar V, Lyons J, Bottomley I, McCaul D, Clarke NW, Kiltie AE, Cowan RA. Phase II study of conformal hypofractionated radiotherapy with concurrent gemcitabine in muscle-invasive bladder cancer. J Clin Oncol. 2011 Feb 20;29(6):733-8. doi: 10.1200/JCO.2010.31.5721. Epub 2011 Jan 4. PMID 21205754
- [Background] Dunst J, Sauer R, Schrott KM, Kuhn R, Wittekind C, Altendorf-Hofmann A. Organ-sparing treatment of advanced bladder cancer: a 10-year experience. Int J Radiat Oncol Biol Phys. 1994 Sep 30;30(2):261-6. doi: 10.1016/0360-3016(94)90003-5. PMID 7928455
- [Background] Ensign LG, Gehan EA, Kamen DS, Thall PF. An optimal three-stage design for phase II clinical trials. Stat Med. 1994 Sep 15;13(17):1727-36. doi: 10.1002/sim.4780131704. PMID 7997706
- [Background] Fechner G, Perabo FG, Schmidt DH, Haase L, Ludwig E, Schueller H, Blatter J, Mller SC, Albers P. Preclinical evaluation of a radiosensitizing effect of gemcitabine in p53 mutant and p53 wild type bladder cancer cells. Urology. 2003 Feb;61(2):468-73. doi: 10.1016/s0090-4295(02)02156-8. PMID 12597983
- [Background] Hagan MP, Winter KA, Kaufman DS, Wajsman Z, Zietman AL, Heney NM, Toonkel LM, Jones CU, Roberts JD, Shipley WU. RTOG 97-06: initial report of a phase I-II trial of selective bladder conservation using TURBT, twice-daily accelerated irradiation sensitized with cisplatin, and adjuvant MCV combination chemotherapy. Int J Radiat Oncol Biol Phys. 2003 Nov 1;57(3):665-72. doi: 10.1016/s0360-3016(03)00718-1. PMID 14529770
- [Background] Herman JM, Smith DC, Montie J, Hayman JA, Sullivan MA, Kent E, Griffith KA, Esper P, Sandler HM. Prospective quality-of-life assessment in patients receiving concurrent gemcitabine and radiotherapy as a bladder preservation strategy. Urology. 2004 Jul;64(1):69-73. doi: 10.1016/j.urology.2004.02.024. PMID 15245938
- [Background] Housset M, Maulard C, Chretien Y, Dufour B, Delanian S, Huart J, Colardelle F, Brunel P, Baillet F. Combined radiation and chemotherapy for invasive transitional-cell carcinoma of the bladder: a prospective study. J Clin Oncol. 1993 Nov;11(11):2150-7. doi: 10.1200/JCO.1993.11.11.2150. PMID 8229129
- [Background] Kent E, Sandler H, Montie J, Lee C, Herman J, Esper P, Fardig J, Smith DC. Combined-modality therapy with gemcitabine and radiotherapy as a bladder preservation strategy: results of a phase I trial. J Clin Oncol. 2004 Jul 1;22(13):2540-5. doi: 10.1200/JCO.2004.10.070. PMID 15226322
- [Background] Lagrange JL, Bascoul-Mollevi C, Geoffrois L, Beckendorf V, Ferrero JM, Joly F, Allouache N, Bachaud JM, Chevreau C, Kramar A, Chauvet B; Study Group on Genito-Urinary Tumors. Quality of life assessment after concurrent chemoradiation for invasive bladder cancer: results of a multicenter prospective study (GETUG 97-015). Int J Radiat Oncol Biol Phys. 2011 Jan 1;79(1):172-8. doi: 10.1016/j.ijrobp.2009.10.038. Epub 2010 Apr 10. PMID 20385453
- [Background] Lawrence TS, Chang EY, Hahn TM, Shewach DS. Delayed radiosensitization of human colon carcinoma cells after a brief exposure to 2',2'-difluoro-2'-deoxycytidine (Gemcitabine). Clin Cancer Res. 1997 May;3(5):777-82. PMID 9815749
- [Background] Moore MJ, Tannock IF, Ernst DS, Huan S, Murray N. Gemcitabine: a promising new agent in the treatment of advanced urothelial cancer. J Clin Oncol. 1997 Dec;15(12):3441-5. doi: 10.1200/JCO.1997.15.12.3441. PMID 9396395
- [Background] Rodel C, Grabenbauer GG, Kuhn R, Papadopoulos T, Dunst J, Meyer M, Schrott KM, Sauer R. Combined-modality treatment and selective organ preservation in invasive bladder cancer: long-term results. J Clin Oncol. 2002 Jul 15;20(14):3061-71. doi: 10.1200/JCO.2002.11.027. PMID 12118019
- [Background] Sangar VK, McBain CA, Lyons J, Ramani VA, Logue JP, Wylie JP, Clarke NW, Cowan RA. Phase I study of conformal radiotherapy with concurrent gemcitabine in locally advanced bladder cancer. Int J Radiat Oncol Biol Phys. 2005 Feb 1;61(2):420-5. doi: 10.1016/j.ijrobp.2004.05.074. PMID 15667962
- [Background] Shewach DS, Hahn TM, Chang E, Hertel LW, Lawrence TS. Metabolism of 2',2'-difluoro-2'-deoxycytidine and radiation sensitization of human colon carcinoma cells. Cancer Res. 1994 Jun 15;54(12):3218-23. PMID 8205542
- [Background] Shipley WU, Kaufman DS, Tester WJ, Pilepich MV, Sandler HM; Radiation Therapy Oncology Group. Overview of bladder cancer trials in the Radiation Therapy Oncology Group. Cancer. 2003 Apr 15;97(8 Suppl):2115-9. doi: 10.1002/cncr.11282. PMID 12673704
- [Background] Stadler WM, Kuzel T, Roth B, Raghavan D, Dorr FA. Phase II study of single-agent gemcitabine in previously untreated patients with metastatic urothelial cancer. J Clin Oncol. 1997 Nov;15(11):3394-8. doi: 10.1200/JCO.1997.15.11.3394. PMID 9363871
- [Background] Stein JP, Lieskovsky G, Cote R, Groshen S, Feng AC, Boyd S, Skinner E, Bochner B, Thangathurai D, Mikhail M, Raghavan D, Skinner DG. Radical cystectomy in the treatment of invasive bladder cancer: long-term results in 1,054 patients. J Clin Oncol. 2001 Feb 1;19(3):666-75. doi: 10.1200/JCO.2001.19.3.666. PMID 11157016
- [Background] Tester W, Caplan R, Heaney J, Venner P, Whittington R, Byhardt R, True L, Shipley W. Neoadjuvant combined modality program with selective organ preservation for invasive bladder cancer: results of Radiation Therapy Oncology Group phase II trial 8802. J Clin Oncol. 1996 Jan;14(1):119-26. doi: 10.1200/JCO.1996.14.1.119. PMID 8558186
- [Background] Advanced Bladder Cancer Meta-analysis Collaboration. Neoadjuvant chemotherapy in invasive bladder cancer: a systematic review and meta-analysis. Lancet. 2003 Jun 7;361(9373):1927-34. doi: 10.1016/s0140-6736(03)13580-5. PMID 12801735
- [Background] Vogelzang NJ, Stadler WM. Gemcitabine and other new chemotherapeutic agents for the treatment of metastatic bladder cancer. Urology. 1999 Feb;53(2):243-50. doi: 10.1016/s0090-4295(98)00501-9. PMID 9933034
- [Background] von der Maase H, Hansen SW, Roberts JT, Dogliotti L, Oliver T, Moore MJ, Bodrogi I, Albers P, Knuth A, Lippert CM, Kerbrat P, Sanchez Rovira P, Wersall P, Cleall SP, Roychowdhury DF, Tomlin I, Visseren-Grul CM, Conte PF. Gemcitabine and cisplatin versus methotrexate, vinblastine, doxorubicin, and cisplatin in advanced or metastatic bladder cancer: results of a large, randomized, multinational, multicenter, phase III study. J Clin Oncol. 2000 Sep;18(17):3068-77. doi: 10.1200/JCO.2000.18.17.3068. PMID 11001674
- [Derived] Azria D, Riou O, Rebillard X, Thezenas S, Thuret R, Fenoglietto P, Pouessel D, Culine S. Combined chemoradiation therapy with twice-weekly gemcitabine and cisplatin for organ preservation in muscle-invasive bladder cancer: long-term results of a phase 1 trial. Int J Radiat Oncol Biol Phys. 2014 Mar 15;88(4):853-9. doi: 10.1016/j.ijrobp.2013.11.016. Epub 2013 Dec 21. PMID 24368064

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiotherapy + Cisplatin | Radiotherapy + Cisplatin + Gemcitabine
Started | 24 | 45
Completed | 24 | 43
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiotherapy + Cisplatin | Radiotherapy + Cisplatin + Gemcitabine | Total
Number analyzed (Participants) | 24 | 45 | 69
Age, Continuous [Median (Full Range); unit: years] | 76.5 [57 to 84] | 71 [54 to 86] | 72 [54 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 22 | 39 | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: The time to relapse is defined as the time from the date of randomisation to the date of the first event. Time to relapse for patients without any event (local, regional, distance, or death) will be censored at the date of latest information.
  Patients without relapse and living at 2 years will be considered a success
Time Frame: Two years after the end of the complete therapeutic sequence
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy + Cisplatin | Radiotherapy + Cisplatin + Gemcitabine
Number analyzed (Participants) | 24 | 45
Participants
  Number of patients without any event (local, regional, distance, or death) | 11 | 22
  Number of patients with any event (local, regional, distance, or death) | 13 | 23

2. Secondary Outcome: Overall Survival
Description: The time to death is defined as time from the randomization to the date of death from any cause, or to the date on which latest information is obtained.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy + Cisplatin | Radiotherapy + Cisplatin + Gemcitabine
Number analyzed (Participants) | 24 | 45
Participants
  number of patient alive | 17 | 25
  number of patient death | 7 | 20

3. Secondary Outcome: Acute and Late Toxicities
Description: Acute and late toxicities will be scored according to the NCI-CTC v4.0. Grade 0 : no toxicity Grade 4 : worse toxicity
Time Frame: Up to 5 years
Population: Analyses are performed on the population that can be evaluated for tolerance
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy + Cisplatin | Radiotherapy + Cisplatin + Gemcitabine
Number analyzed (Participants) | 24 | 43
Participants
  late toxicity per patient: grade < 3 | 21 | 40
  late toxicity per patient: grade 3/4 | 3 | 3
  acute toxicity per patient: grade < 3 | 21 | 20
  acute toxicity per patient: grade 3/4 | 3 | 23

4. Secondary Outcome: Correlation Between Lymphocyte Apoptosis and Severity of Late Toxicities.
Description: Before starting radiotherapy, 5ml of blood will be sampled in a 5ml heparinised tube to prospectively measure the rate of CD8 radio-induced lymphocyte apoptosis before any radiotherapy treatment. A correlation between the low rate of lymphocyte apoptosis and the severity of late toxicities will be studied to confirm the predictive power of this biological test on radio-induced side-effects.
  Percentage of Cell Death Measured by Apoptosis This Outcome Measure was pre-specified to report based on toxicity event instead of assigned intervention
Time Frame: Up to 5 years
Population: patient groups were defined in order to validate a possible correlation between the apoptosis rate observed during blood analysis and the severe toxicity rate.
Measure: Mean (Standard Deviation); unit: Percentage of dead Cells
Groups:
- Patients Without Severe Toxicity (Acute and Late): no toxicity
- Patients Without Severe Acute Toxicity: patient with acute severe toxicity
- Patients Without Severe Late Toxicity: patient with late severe toxicity
- Patients With Severe Toxicity (Acute and Late): patient with acute and late severe toxicity
Arm/Group | Patients Without Severe Toxicity (Acute and Late) | Patients Without Severe Acute Toxicity | Patients Without Severe Late Toxicity | Patients With Severe Toxicity (Acute and Late)
Number analyzed (Participants) | 7 | 10 | 2 | 2
Percentage of dead Cells
  Apoptosis CD8 spontaneous | 2.9 (1.4) | 2.7 (1.4) | 3.4 (1.4) | 2.9 (0.4)
  Apoptosis CD8 to 8 Gy | 20.9 (11.6) | 30.9 (16.6) | 28.3 (13.4) | 26.3 (6.4)
  Radio-induced CD8 apoptosis | 18 (10.7) | 28.2 (15.91) | 24.9 (11.9) | 23.4 (6)

ADVERSE EVENTS:
Time Frame: collection from the baseline to 5 years afetr the treatment
Description: Analyses are performed on the population assessable for tolerance, 24 vs 43 pts in the arms RT/CDDP and RT/CDDP/GEMZAR; Two pts RT/CDDP/GEMAZR having not treated.
  only toxicities are discussed in Probable/Possible relationship with treatment. All patients reported at least toxicity. Two patients showed no toxicity his Outcome Measure was pre-specified to report based on toxicity event instead of assigned intervention", or similar, as accurate and appropriate
Arm/Group | Radiotherapy + Cisplatin | Radiotherapy + Cisplatin + Gemcitabine
All-Cause Mortality (participants affected / at risk) | 7/24 | 20/45
Serious Adverse Events (participants affected / at risk) | 9/24 | 23/45
Other Adverse Events (participants affected / at risk) | 24/24 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiotherapy + Cisplatin (N=24) | Radiotherapy + Cisplatin + Gemcitabine (N=45)
thrombopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
large instestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
small instestinal obtstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
asthenia (General disorders) | 0 (0) | 1 (1)
radiation proctitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
gastroenteritis radiation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
sepsis (Infections and infestations) | 0 (0) | 1 (1)
acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
hematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
atrial flutter (Cardiac disorders) | 0 (0) | 2 (2)
streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiotherapy + Cisplatin (N=24) | Radiotherapy + Cisplatin + Gemcitabine (N=45)
alopecia (General disorders) | 0 (0) | 1 (1) — grade 2
anorexia (Gastrointestinal disorders) | 1 (1) | 14 (14) — Grade 1 to 3
Asthenia (General disorders) | 15 (15) | 27 (27) — grade 1 to 3
Other toxicity (General disorders) | 20 (20) | 40 (40) — grade 1 to 4
Diarrhea (Gastrointestinal disorders) | 13 (13) | 25 (25) — grade 1 to 3
abdominal pain (Gastrointestinal disorders) | 3 (3) | 12 (12) — grade 1 and 2
dysgueusia (General disorders) | 1 (1) | 4 (4) — grade 1 and 2
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — grade 1
dysuria (Renal and urinary disorders) | 6 (6) | 16 (16) — grade 1 and 2
fever (Infections and infestations) | 0 (0) | 3 (3) — grade 1 to 4
hematuria (Renal and urinary disorders) | 5 (5) | 5 (5) — grade 1 to 3
infection (Infections and infestations) | 0 (0) | 2 (2) — grade 2 and 4
urinary infection (Infections and infestations) | 14 (14) | 24 (24) — grade 1 and 2
mucocitis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) — grade 1
nausea (Gastrointestinal disorders) | 8 (8) | 23 (23) — grade 1 and 2
neuropathy (Nervous system disorders) | 1 (1) | 2 (2) — grade 1
pollakiuria (Renal and urinary disorders) | 17 (17) | 26 (26) — grade 1 to 3
audition toxicity (Ear and labyrinth disorders) | 1 (1) | 3 (3) — grade 1 and 2
vomiting (Gastrointestinal disorders) | 3 (3) | 5 (5) — grade 1 and 2

LIMITATIONS AND CAVEATS:
no data for Measurement of Quality of Life

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT01495676/Prot_SAP_000.pdf